CLINICAL TRIAL: NCT04812899
Title: Implementation of a Waitlist Intervention and Clinical Care Pathway for Families Awaiting Services at McMaster Children's Hospital Eating Disorders Program: A Feasibility Study
Brief Title: Implementation of a Waitlist Intervention and Clinical Care Pathway for Families Awaiting at Eating Disorders Program
Acronym: WICFAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Jennifer Couturier, Principal Investigator, McMaster University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 13223
Record Dates: First submitted 2021-03-18; First posted 2021-03-24 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Eating Disorders
Keywords: eating disorders; waitlist intervention; pandemic; children; clinical care pathway
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parents who have a child/adolescent with an eating disorder on waitlist (Experimental): Each participant will receive a series of pre-recorded videos and book -(10 videos of about 10 minutes each, along with the book "Help Your Teenager Beat an Eating Disorder"). This will include content on empowering parents to renourish their child and interrupt binge/purge behaviors.
  Interventions: Behavioral: Parental guided self-help version of FBT-pre-recorded videos and readings from the book

INTERVENTIONS:
Behavioral: Parental guided self-help version of FBT-pre-recorded videos and readings from the book — Each participant will receive a series of pre-recorded videos of parental guided self help version FBT. There will be10 videos of about 10 minutes each. The videos will include content on empowering parents to renourish their child and interrupt binge/purge behaviors. Readings will be assigned to each participant from the book "Help Your Teenager Beat and Eating Disorder". There will be psychoeducational content on the dangers and medical complications of eating disorders. The readings will also contain content on coping skills for young people including relaxation, mindfulness strategies, and distress tolerance skills.

SUMMARY:
The COVID-19 pandemic has resulted in several challenges in service delivery for the eating disorders program at McMaster Children's Hospital. Long waiting lists prior to the pandemic (6-9 month wait time) have been made worse by an interruption in service during the initial stages of the pandemic. New routine assessments were placed on hold for many months, while only the most urgently ill children were seen. This, in combination with a dramatic increase in new referrals has resulted in a long waitlist. Now families are waiting 12-18 months for service. The resulting waitlist is now unmanageable and unsafe. Investigators wish to study the implementation of a waitlist intervention which will educate parents on how to start to renourish their children and interrupt eating disordered behaviors. The intervention will consist of a series of educational videos and a book on how to help their children. It is hoped that this intervention can lessen the need for hospitalization and can change the trajectory of symptoms while waiting for service. A clinical care pathway will also be developed to ensure those waiting receive the most appropriate treatment.

DETAILED DESCRIPTION:
Investigators would like to study the implementation of an adapted FBT model in which there is no therapist involvement and the intervention is delivered to families on the waitlist of Eating Disorder program at McMaster Children's Hospital. The intervention would involve a series of prerecorded videos and reading material. This, in combination with the development of a clinical care pathway, would help to manage the extraordinary volumes of referrals recently been received. The need to social distance brought on by the pandemic presents the opportunity to consider the value of this waitlist intervention as a structured program for parents who have a child waiting for service. A model such as this could dramatically improve parental abilities to begin to re-feed their children, thereby reducing acuity and time spent in treatment. Similarly, some parents on the waitlist may decide that the proposed treatment model is not suitable after they have received the proposed waitlist intervention, and may wish to seek treatment elsewhere. Alternatively, parents may be able to shift the pattern of weight loss and/or binge purge behavior in children so that the severity of illness is decreased by the time of assessment. If successful, this intervention and clinical care pathway for waitlisted patients and their families could be disseminated to other tertiary care centers, thereby reducing mounting pressures on these centers.

ELIGIBILITY:
Inclusion Criteria:

1. Parents of a child or adolescent (6-17 years) with an Eating Disorder.
2. Have an access to the internet/computer.
3. Have an access to a weigh scale in their home environment
4. Have the capacity to write, speak and understand English

Exclusion Criteria:

1. don't have the capacity to write, speak and understand English
2. don't have access to the internet/computer
3. don't have a child or adolescent with an eating disorder

Ages: 7 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-02-04 (Actual)

PRIMARY OUTCOMES:
Weight trajectory | Weight will be collected weekly (in kgs) for 14 weeks. (6 weeks pre intervention, 2 weeks during intervention and 6 weeks post intervention)
  Change in weight trajectory will be measured over the time period of 14 weeks, starting from the Baseline till the end of the study at 14 weeks
Binge/purge episodes trajectory | Number of binge/purge episodes will be collected weekly for 14 weeks. (6 weeks pre intervention, 2 weeks during intervention and 6 weeks post intervention)
  Change in trajectory of symptoms (number of binge/purge episodes) will be measured pre and post intervention.
Length of wait time | At 14 weeks
  Average length of wait time pre and post implementation will be determined by examining wait time in the month prior to implementation for new referrals, compared to the average wait time for new referrals in the month following the completion of the study period
Change in number of parents who accepted to participate in the study | Baseline and at 14 weeks
  In terms of recruitment, the investigators will examine the number of parents agree to participate versus the number of families invited to the study.
Change in number of parents who remain in the study | Baseline and at 14 weeks
  In terms of retention, the investigators will compare the number of parents completed the study to the number of parents enrolled.

SECONDARY OUTCOMES:
Change in Eating Disorder Questionnaire -parent version | Baseline and at 14 weeks
  Eating Disorder Examination Questionnaire -parent version (EDE-Q) will measures the severity of the characteristic psychopathology of eating disorders. The EDE-Q yields four subscale scores (Restraint, Eating Concern, Weight Concern, and Shape Concern) and a global score measuring the overall severity of eating disorder psychopathology.
Change in Parent Versus Eating Disorder Scale | Baseline and at 14 weeks
  Parent Versus Eating Disorder Scale (PvEDs) is a self-efficacy tool, specifically focused on parental self-efficacy related to re-feeding their child with an Eating Disorder.
Change in Nine Item Avoidant/Restrictive Food Intake disorder screen | Baseline and at 14 weeks
  Nine Item Avoidant/Restrictive Food Intake disorder screen (NIAS) -Parental version is a 9-item, Likert scale questionnaire that inquires about picky eating, interest in food, and eating habits driven by a fear of negative consequences. Minimum score is 0 and maximum is 45. A score of ≥ 24 is considered a positive ARFID screen.
Change in Pediatric Symptom Checklist-17 | Baseline and at 14 weeks
  Pediatric Symptom Checklist-17 (PSC-17) is a 17-item general mental health screening tool that can help to assess the likelihood of finding any mental health disorder. Minimum score is 0 and maximum is 35. A total score of 15 or more points may indicate the need for a referral to a qualified medical or mental health professional.
Change in Carers Needs Assessment Measure | Baseline and at 14 weeks
  Carers Needs Assessment Measure (CaNAM): This 47 item questionnaire is designed to assess the needs of a carer of someone with an eating disorder. The minimum score is 0, the maximum score is 64. A higher score indicates that the carer has received sufficient information and support for themselves and their child.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Couturier, MD, Principal Investigator — McMaster University
Locations (1):
- McMaster Children's Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No